CLINICAL TRIAL: NCT05826717
Title: Effects of the Food Matrix on Serum Fructose Peaks
Brief Title: Effect of Matrices on Serum Fructose.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NL81668.068.22
Record Dates: First submitted 2023-03-28; First posted 2023-04-24 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Fructose Metabolism Disorder
MeSH Terms: interventions — Water

STUDY DESIGN:
Intervention Model Description: This study is an open-label, randomized, single meal, cross-over study in healthy individuals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Food product 1. (Experimental): [x] gr apple containing 20 gr fructose as measured with an enzymatic method. Administered one time.
  Interventions: Other: Apple
- Food product 2. (Experimental): [x] gr mashed apple containing 20 gr fructose as measured with an enzymatic method. Administered one time.
- Food product 3. (Experimental): [x] ml apple juice containing 20 gr fructose as measured with an enzymatic method. Administered one time.
  Interventions: Other: Apple juice
- Food product 4. (Experimental): 20 gr of fructose powder dissolved in 300 ml of water. Administered one time.
  Interventions: Other: Fructose powder in water

INTERVENTIONS:
Other: Apple — 20g fructose in [x] g of apple
  Arms: Food product 1.
Other: Mashed apple — 20g fructose in [x] g of mashed apple
Other: Apple juice — 20g fructose in [x] ml apple juice
  Arms: Food product 3.
Other: Fructose powder in water — 20g fructose in [x] ml water
  Arms: Food product 4.

SUMMARY:
Epidemiological evidence is accumulating that a high consumption of added sugars is associated with metabolic diseases such as non-alcoholic fatty liver disease and type 2 diabetes. Fructose, one of the principal added sugars, is believed to be the most disadvantageous sugar. Data from a large population-based cohort demonstrated that fructose intake from fruit juice and sugar-sweetened beverages, but not whole fruits, is associated with higher intrahepatic lipid content. A study in mice demonstrated that fast fructose exposure resulted in higher intrahepatic lipid content than slow fructose exposure.

The food matrix, i.e. the complex spatial organisation of and interactions between nutrients, may account for the fast versus slow fructose exposure and subsequent health consequences. Therefore the investigators aim to investigate the role of the fructose matrices on serum fructose peaks. The investigators hypothesize that liquid fructose matrices will cause higher serum fructose peaks in comparison to solid fructose matrices.

Objective: To quantify serum fructose peaks within 150 minutes following intake of fructose-containing matrices.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Body mass index (BMI) ≥18.5 kg/m2 and <25 kg/m2

Exclusion Criteria:

* Pregnancy.
* Drugs and/or alcohol abuse.
* Diagnosis of diabetes mellitus.
* (History of) gastrointestinal and/or liver disease.
* (History [< 5 years] of) cancer (excluding basal cell carcinoma)
* Physical stress one month prior to inclusion (i.e. post-surgery, trauma that requires medical treatment, bacterial/viral/fungal infection or extreme psychological stress). Symptoms of infection include: fever, (excessive) sweating & chills, cough, sore throat, shortness of breath, nasal congestion, diarrhea, vomiting, painful miction, redness/swelling, stomach ache, head ache, and stiff neck.
* Unstable weight for 3 months prior to inclusion (i.e. 5% change in bodyweight)
* Allergy to one of the used food products in the study.
* Inability to provide written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Change in serum fructose between peak and baseline | Time points 0, 15, 30, 45, 60, 75, 90, 105, 120, 135 and 150 minutes following consumption of the food product.

SECONDARY OUTCOMES:
Blood pressure | Time points 0, 15, 30, 45, 60, 75, 90, 105, 120, 135 and 150 minutes following consumption of the food product.
  Millimeter of mercury
Serum uric acid | Time points 0, 15, 30, 45, 60, 75, 90, 105, 120, 135 and 150 minutes following consumption of the food product.
  Millimoles per liter

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Hospital Maastricht, Maastricht, Netherlands